CLINICAL TRIAL: NCT00349544
Title: Validation of the Transcultural Adaptation of the Neck Disability Index in the Spanish Population
Brief Title: Validation of the Spanish Version of the Neck Disability Index
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Collaborators: Spanish Back Pain Research Network (REIDE) (Other)
Responsible Party: Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation
Other Study IDs: FK-R-10
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Neck Pain; Cervicalgia
Keywords: Neck pain; Cervicalgia; Quality of life; Disability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to adapt the Neck Disability Index (NDI)and the Cervical Core Set 6 (CCS6) to the Spanish population. Other objectives are to determine the correlation between intensity of cervical pain, degree of disability, and quality of life; to determine the correlation between the NDI, CCS6 and the Northwick Park Neck Pain Questionnaire; and to determine factors that predict the chronification of disability.

ELIGIBILITY:
Inclusion Criteria:

* patients who visit physician for cervicalgia
* with or without referred pain
* must be able to read and write

Exclusion Criteria:

* disease of central nervous system, with or without treatment
* migraine
* indications for surgery
* suspicion of systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit their physician for cervicalgia, with or without referred pain
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2005-10; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M. Kovacs, MD, PhD, Study Chair — Kovacs Foundation, Palma de Mallorca 07012, Spain; Juan Bago, MD, Study Director — Hospital Vall d'Hebron 119-129, Barcelona 08035, Spain; Luis Cuesta, MD, Study Director — Mutua Asepeyo, Madrid 28820, Spain; José Luis Martín, MD, Study Director — Hospital Universitario Virgen de las Nieves, Granada 18014, Spain; Luis Alvarez, MD, Study Director — Fundación Jiménez Díaz, Madrid 28040, Spain; María Angeles Usero, MD, Study Director — Centro de Salud Perales del Rio, Madrid 28909, Spain; Carmen Fernández, MD, Study Director — Centro de Salut de Valldargent, Palma de Mallorca 07013, Spain; María Dolores Castillo, MD, Study Director — Delegación Pral. de Asuntos Sociales, Granada 18011, Spain; Montserrat Cañellas, MD, Study Director — Consorci Sanitari del Parc Taulí, Hospital Sabadell, Barcelona 08208, Spain; Montserrat Núñez, MD, Study Director — Hospital Clínic de Barcelona, Barcelona 08036, Spain; Sergio Giménez, MD, Study Director — Centro de Salud Ciudad Jardín, Málaga 29017, Spain; Pablo Panero, MD, Study Director — ZBS Órgiva, Granada 18640, Spain; Luis González, MD, Study Director — Centro de Salud Serrería II, Valencia 46022, Spain; Myriam Bernal, MD, Study Director — Servicio de Rehabilitación del Hospital Clínico de Valladolid, Valladolid 47002, Spain; Mateo Seguí, MD, Study Director — Unidad Básica de Salut Es Castell, Menorca 07720, Spain; Víctor Abraira, PhD, Study Director — Unidad de Bioestadística, Hospital Ramón y Cajal, Madrid 28034, Spain
Locations (1):
- Fundación Kovacs, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Derived] Kovacs FM, Bago J, Royuela A, Seco J, Gimenez S, Muriel A, Abraira V, Martin JL, Pena JL, Gestoso M, Mufraggi N, Nunez M, Corcoll J, Gomez-Ochoa I, Ramirez MJ, Calvo E, Castillo MD, Marti D, Fuster S, Fernandez C, Gimeno N, Carballo A, Milan A, Vazquez D, Canellas M, Blanco R, Brieva P, Rueda MT, Alvarez L, Del Real MT, Ayerbe J, Gonzalez L, Ginel L, Ortega M, Bernal M, Bolado G, Vidal A, Ausin A, Ramon D, Mir MA, Tomas M, Zamora J, Cano A. Psychometric characteristics of the Spanish version of instruments to measure neck pain disability. BMC Musculoskelet Disord. 2008 Apr 9;9:42. doi: 10.1186/1471-2474-9-42. PMID 18400084
- See also: Spanish Back Pain Research Network site that describes objectives and projects of its members. — http://www.reide.org